CLINICAL TRIAL: NCT02070718
Title: Effects of a Kappa Agonist on Hot Flashes in Menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Research on Women's Health (ORWH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Susan Reed, Professor, Obstetrics & Gynecology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43952-B; GYN-01-2012 (Other: University of Washington)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Treatment of Menopausal Hot Flashes
Keywords: hot flashes; menopause; kappa agonist
MeSH Terms: conditions — Hot Flashes | interventions — Pentazocine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Cornstarch, National Formulary
  Interventions: Other: Placebo
- Standard Dose Kappa Agonist (Experimental): Pentazocine/Naloxone 50/0.5 mg
  Interventions: Drug: Standard Dose Kappa Agonist
- Half Dose Kappa Agonist (Experimental): Pentazocine/Naloxone 25/0.25 mg
  Interventions: Drug: Half Dose Kappa Agonist

INTERVENTIONS:
Drug: Standard Dose Kappa Agonist
  Other Names: Pentazocine/Naloxone 50/0.5 mg
  Arms: Standard Dose Kappa Agonist
Drug: Half Dose Kappa Agonist
  Other Names: Pentazocine/Naloxone 25/0.25 mg
  Arms: Half Dose Kappa Agonist
Other: Placebo
  Arms: Placebo

SUMMARY:
Studies suggest that kappa agonists (KA) and peripherally restricted kappa agonists (PRKAs) may affect thermoregulation. This pilot study has the aim to establish proof of concept regarding efficacy of an oral kappa agonist (KA) for the treatment of menopausal hot flashes.

DETAILED DESCRIPTION:
To establish proof of concept regarding efficacy of an oral kappa agonist (KA), Pentazocine/ Naloxone 50/0.5 mg, for the treatment of menopausal hot flashes.

To gather data in support of a future proposal to study the safety and efficacy of a PRKA, a type of KA, for amelioration of menopausal hot flashes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women 45-60 years of age; 12 months amenorrhea
2. Documentation of > 8 moderate to severe, daily hot flashes during one week of baseline monitoring using daily diaries
3. Availability of a family member or friend to drive participant home following clinic visits

Exclusion Criteria:

1. Use of hormonal prescription medication or supplements for vasomotor symptoms (VMS)
2. Use of narcotics
3. Use of SSRI (selective serotonin reuptake inhibitor)/SNRI (serotonin-norepinephrine reuptake inhibitors), gabapentin, MAOI (monoamine oxidase inhibitor), anti-epileptics, sedatives
4. History of polycystic ovarian syndrome or hirsutism
5. Current history of depression
6. Any chronic or acute medical illnesses including renal, hepatic, pulmonary diseases, or seizures
7. Substance abuse
8. Severe corn allergy
9. Known allergic reaction to pentazocine or naloxone
10. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
11. Hysterectomy
12. Use of anticholinergic medications
13. Lactating or pregnant

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Hot Flashes | 1-4 weeks
  Objectively measured hot flash frequency by changes in skin conductance over 8 hours on 3 separate study visits 3-14 days apart.

SECONDARY OUTCOMES:
Subjectively measured hot flashes | 1-4 weeks
  Self-reported diary documentation of time and occurence of hot flashes and intensity of hot flashes over 8 hours on 3 separate study visits 3-14 days apart.
Change in Serum Leutinizing Hormone | 1-4 weeks
  Serum collected at each visit baseline (before administration of treatment) and at 20-minute intervals over 8 hours on 3 separate study visits 3-14 days apart.

OTHER OUTCOMES:
Serum Follicle Stimulating Hormone | Baseline only
  Baseline (1st visit) single time point
Serum Estradiol | Baseline only
  Baseline (1st visit) single time point only.

CONTACTS AND LOCATIONS:
Overall Officials: Susan D Reed, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Oakley AE, Steiner RA, Chavkin C, Clifton DK, Ferrara LK, Reed SD. kappa Agonists as a novel therapy for menopausal hot flashes. Menopause. 2015 Dec;22(12):1328-34. doi: 10.1097/GME.0000000000000476. PMID 25988798